CLINICAL TRIAL: NCT05171855
Title: A Multicenter, Open-Label, Extension Trial to Investigate Long Term Efficacy and Safety of Lonapegsomatropin in Adults With Growth Hormone Deficiency
Brief Title: A Trial to Investigate Long Term Efficacy and Safety of Lonapegsomatropin in Adults With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma Endocrinology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCH-306EXT
Record Dates: First submitted 2021-09-24; First posted 2021-12-29 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Adult Growth Hormone Deficiency; Endocrine System Diseases; Hormone Deficiency
Keywords: Human Growth Hormone; hGH; rhGH; GHD; Adult Growth Hormone Deficiency; Long Acting Growth Hormone; Lonapegsomatropin; Prodrug; Growth Hormone Replacement Therapy; Sustained Release Growth Hormone; Growth Hormone Deficiency; TransCon hGH; Skytrofa
MeSH Terms: conditions — Dwarfism, Pituitary; Endocrine System Diseases | interventions — lonapegsomatropin

STUDY DESIGN:
Intervention Model Description: Open label treatment with weekly Lonapegsomatropin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lonapegsomatropin/Lonapegsomatropin (Experimental): Participants who had completed treatment with lonapegsomatropin in TCH-306 study were enrolled in the extension study and received lonapegsomatropin administered once weekly by subcutaneous injection for a treatment period of up to 52 weeks.
  Interventions: Drug: Lonapegsomatropin
- Placebo/Lonapegsomatropin (Experimental): Participants who had completed treatment with placebo in TCH-306 study were enrolled in the extension study and received lonapegsomatropin administered once weekly by subcutaneous injection for a treatment period of up to 52 weeks.
  Interventions: Drug: Lonapegsomatropin
- Somatropin/Lonapegsomatropin (Experimental): Participants who had completed treatment with somatropin in TCH-306 study were enrolled in the extension study and received lonapegsomatropin administered once weekly by subcutaneous injection for a treatment period of up to 52 weeks.
  Interventions: Drug: Lonapegsomatropin

INTERVENTIONS:
Drug: Lonapegsomatropin — Study participants were individually dosed with subcutaneous injection of Lonapegsomatropin once-weekly for 52 weeks.
  Other Names: ACP-011

SUMMARY:
This was a phase 3 open-label multicenter extension study designed to evaluate the long-term safety and efficacy of Lonapegsomatropin administered once-weekly. The study participants were adults (males and females) with confirmed growth hormone deficiency (GHD) having completed the treatment period in study TCH-306 (foresiGHt; NCT04615273).

ELIGIBILITY:
Inclusion Criteria:

* Signing of the trial specific informed consent
* Completion of the treatment period and Visit 7 assessments of trial TCH-306, including collection and upload of Visit 7 dual-X-ray-absorptiometry (DXA) scan
* Fundoscopy at Visit 7 in trial TCH-306 without signs/symptoms of intracranial hypertension or diabetic retinopathy stage 2 / moderate or above

Exclusion Criteria:

* Diabetes mellitus if any of the following were met:

  1. Poorly controlled diabetes, defined as HbA1C higher than 7.5% according to central laboratory at Visit 7 in trial TCH-306
  2. Use of diabetes mellitus drugs other than metformin and/or dipeptidyl peptidase-4 (DPP-4) inhibitors
* Active malignant disease or history of malignancy.
* Known history of hypersensitivity and/or idiosyncrasy to the investigational product (somatropin or excipients)
* Female who was pregnant, plans to become pregnant, or was breastfeeding
* Female participant of childbearing potential (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile) not willing throughout the trial to use contraceptives as required by local law or practice. Details included in Appendix 4/section 10.4 of the protocol
* Male participant not willing throughout the trial to use contraceptives as required by local law or practice. Details included in Appendix 4/ section 10.4 of the protocol
* Any disease or condition that, in the judgement of the investigator, may make the participant unlikely to comply with the requirements of the protocol or any condition that presents undue risk from the investigational product or trial procedures

Ages: 23 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Strange, Study Director — Ascendis Pharma A/S
Locations (79):
- United States (15):
  - Ascendis Pharma Investigational Site, Phoenix, Arizona
  - Ascendis Pharma Investigational Site, Torrance, California
  - Ascendis Pharma Investigational Site, Chicago, Illinois
  - Ascendis Pharma Investigational Site, Indianapolis, Indiana
  - Ascendis Pharma Investigational Site, Boston, Massachusetts
  - Ascendis Pharma Investigational Site, Dearborn, Michigan
  - Ascendis Pharma Investigational Site, Rochester, Minnesota
  - Ascendis Pharma Investigational Site, St Louis, Missouri
  - Ascendis Pharma Investigational Site, Las Vegas, Nevada
  - Ascendis Pharma Investigational Site, Reno, Nevada
  - Ascendis Pharma Investigational Site, New York, New York
  - Ascendis Pharma Investigational Site, Portland, Oregon
  - Ascendis Pharma Investigational Site, Dallas, Texas
  - Ascendis Pharma Investigational Site, San Antonio, Texas
  - Ascendis Pharma Investigational Site, Seattle, Washington
- Ascendis Pharma Investigational Site, Yerevan, Armenia
- Australia (6):
  - Ascendis Pharma Investigational Site, Saint Leonards, New South Wales
  - Ascendis Pharma Investigational Site, Sydney, New South Wales
  - Ascendis Pharma Investigational Site, Box Hill, Victoria
  - Ascendis Pharma Investigational Site, Fitzroy, Victoria
  - Ascendis Pharma Investigational Site, Parkville, Victoria
  - Ascendis Pharma Investigational Site, Perth, Western Australia
- Ascendis Pharma Investigational Site, Halifax, Nova Scotia, Canada
- France (3):
  - Ascendis Pharma Investigational Site, Lyon
  - Ascendis Pharma Investigational Site, Marseille
  - Ascendis Pharma Investigational Site, Nantes
- Ascendis Pharma Investigational Site, Tbilisi, Georgia
- Ascendis Pharma Investigational Site, München, Germany
- Greece (2):
  - Ascendis Pharma Investigational Site, Athens
  - Ascendis Pharma Investigational Site, Thessaloniki
- Israel (3):
  - Ascendis Pharma Investigational Site, Haifa
  - Ascendis Pharma Investigational Site, Petah Tikva
  - Ascendis Pharma Investigational Site, Tel Aviv
- Italy (2):
  - Ascendis Pharma Investigational Site, Genova
  - Ascendis Pharma Investigational Site, Rome
- Japan (19):
  - Ascendis Pharma Investigational Site, Kobe, Hyōgo
  - Ascendis Pharma Investigational Site, Kawasaki, Kanagawa
  - Ascendis Pharma Investigational Site, Yokohama, Kanagawa
  - Ascendis Pharma Investigational Site, Chiba
  - Ascendis Pharma Investigational Site, Fukuoka
  - Ascendis Pharma Investigational Site, Ishikawa
  - Ascendis Pharma Investigational Site, Kagoshima
  - Ascendis Pharma Investigational Site, Kawasaki
  - Ascendis Pharma Investigational Site, Kitakyushu
  - Ascendis Pharma Investigational Site, Matsumoto
  - Ascendis Pharma Investigational Site, Miyakojima
  - Ascendis Pharma Investigational Site, Nagakute
  - Ascendis Pharma Investigational Site, Nara
  - Ascendis Pharma Investigational Site, Okayama
  - Ascendis Pharma Investigational Site, Osaka
  - Ascendis Pharma Investigational Site, Shizuoka
  - Ascendis Pharma Investigational Site, Suita
  - Ascendis Pharma Investigational Site, Yamagata
  - Ascendis Pharma Investigational Site, Yokohama
- Malaysia (3):
  - Ascendis Pharma Investigational Site, George Town
  - Ascendis Pharma Investigational Site, Malacca
  - Ascendis Pharma Investigational Site, Putrajaya
- Poland (4):
  - Ascendis Pharma Investigational Site, Krakow
  - Ascendis Pharma Investigational Site, Lodz
  - Ascendis Pharma Investigational Site, Warsaw
  - Ascendis Pharma Investigational Site, Wroclaw
- Romania (2):
  - Ascendis Pharma Investigational Site, Bucharest
  - Ascendis Pharma Investigational Site, Iași
- Ascendis Pharma Investigational Site, Belgrade, Serbia
- Slovakia (2):
  - Ascendis Pharma Investigational Site, Bratislava
  - Ascendis Pharma Investigational Site, Ľubochňa
- Ascendis Pharma Investigational Site, Soeul, South Korea
- Spain (3):
  - Ascendis Pharma Investigational Site, Alicante
  - Ascendis Pharma Investigational Site, Barcelona
  - Ascendis Pharma Investigational Site, Seville
- Turkey (Türkiye) (5):
  - Ascendis Pharma Investigational Site, Ankara
  - Ascendis Pharma Investigational Site, Antalya
  - Ascendis Pharma Investigational Site, Aydin
  - Ascendis Pharma Investigational Site, İzmit
  - Ascendis Pharma Investigational Site, Kayseri
- Ukraine (3):
  - Ascendis Pharma Investigational Site, Ivano-Frankivsk
  - Ascendis Pharma Investigational Site, Kyiv
  - Ascendis Pharma Investigational Site, Vinnytsia
- Ascendis Pharma Investigational Site, Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study TCH-306 EXT enrolled participants who had completed treatment in TCH-306 (NCT04615273) study. In Japan only, participants switched from commercially available somatropin therapy (results reported separately).
Period: Overall Study
Arm/Group | Lonapegsomatropin/Lonapegsomatropin | Placebo/Lonapegsomatropin | Somatropin/Lonapegsomatropin
Started | 73 | 73 | 74
Completed (Completed 52-Weeks Treatment in TCH-306 EXT) | 67 | 69 | 66
Not Completed | 6 | 4 | 8
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 5
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants who were exposed to any amount of the trial drug in the study TCH-306 EXT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lonapegsomatropin/Lonapegsomatropin | Placebo/Lonapegsomatropin | Somatropin/Lonapegsomatropin | Total
Number analyzed (Participants) | 73 | 73 | 74 | 220
Age, Customized [Count of Participants; unit: Participants]
  < 30 years | 10 | 13 | 14 | 37
  >= 30 to <= 60 years | 53 | 51 | 52 | 156
  > 60 years | 10 | 9 | 8 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 31 | 100
  Male | 36 | 41 | 43 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 5 | 11
  Not Hispanic or Latino | 68 | 69 | 67 | 204
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 9 | 7 | 8 | 24
  Black or African American | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 59 | 62 | 64 | 185
  Other | 5 | 3 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and TEAE Leading to Study Discontinuation
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the treatment. An AE was considered a TEAE if it occurred on or after the first dose of investigational product and was not present prior to the first dose, or it was present at the first dose but increased in severity during the trial. A serious AE was any untoward medical occurrence at any dose that met any of the following criteria: resulted in death; was life threatening; required or prolonged inpatient hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the trial drug or was considered a significant medical event by the investigator.
Time Frame: Up to 52 Weeks
Population: Analysis was performed on all participants who were exposed to any amount of the trial drug in the study TCH-306 EXT.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo/Lonapegsomatropin: Participants who had completed treatment with placebo in TCH-306 study were enrolled in the study and extension study lonapegsomatropin administered once weekly by subcutaneous injection for a treatment period of up to 52 weeks.
Arm/Group | Lonapegsomatropin/Lonapegsomatropin | Placebo/Lonapegsomatropin | Somatropin/Lonapegsomatropin
Number analyzed (Participants) | 73 | 73 | 74
Participants
  TEAEs | 48 | 52 | 45
  Serious TEAEs | 7 | 4 | 5
  TEAE Leading to Study Discontinuation | 2 | 4 | 2

2. Secondary Outcome: Change From Baseline in Trunk Percent Fat at Week 52
Description: Trunk percent fat was assessed by dual-energy X-ray absorptiometry.
Time Frame: Baseline main trial to week 52 (extension period)
Population: Analysis was performed on safety analysis set. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent fat
Arm/Group | Lonapegsomatropin/Lonapegsomatropin | Placebo/Lonapegsomatropin | Somatropin/Lonapegsomatropin
Number analyzed (Participants) | 67 | 69 | 66
percent fat | -1.21 [-2.41 to -0.01] | -1.60 [-2.35 to -0.86] | -1.11 [-2.05 to -0.17]

3. Secondary Outcome: Change From Baseline in Trunk Fat Mass at Week 52
Description: Trunk fat mass was assessed by dual-energy X-ray absorptiometry.
Time Frame: Baseline main trial to week 52 (extension period)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Lonapegsomatropin/Lonapegsomatropin | Placebo/Lonapegsomatropin | Somatropin/Lonapegsomatropin
Number analyzed (Participants) | 67 | 69 | 66
kilograms | 0.15 [-0.47 to 0.77] | -0.16 [-0.63 to 0.31] | -0.00 [-0.53 to 0.53]

4. Secondary Outcome: Change From Baseline in Total Body Lean Mass at Week 52
Description: Total body lean mass was assessed by dual-energy X-ray absorptiometry.
Time Frame: Baseline main trial to week 52 (extension period)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Lonapegsomatropin/Lonapegsomatropin | Placebo/Lonapegsomatropin | Somatropin/Lonapegsomatropin
Number analyzed (Participants) | 67 | 69 | 66
kilograms | 2.26 [1.47 to 3.05] | 1.97 [1.15 to 2.80] | 2.07 [1.21 to 2.94]

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to Week 52
Description: Analysis was performed on all participants who were exposed to any amount of the trial drug in the study TCH-306 EXT.
Arm/Group | Lonapegsomatropin/Lonapegsomatropin | Placebo/Lonapegsomatropin | Somatropin/Lonapegsomatropin
All-Cause Mortality (participants affected / at risk) | 1/73 | 0/73 | 0/74
Serious Adverse Events (participants affected / at risk) | 7/73 | 4/73 | 5/74
Other Adverse Events (participants affected / at risk) | 25/73 | 29/73 | 21/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lonapegsomatropin/Lonapegsomatropin (N=73) | Placebo/Lonapegsomatropin (N=73) | Somatropin/Lonapegsomatropin (N=74)
Sepsis (Infections and infestations) | 2 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Norovirus infection (Infections and infestations) | 1 | 0 | 0
Infected seroma (Infections and infestations) | 0 | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Cerebral cyst (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Sarcoidosis of lymph node (Blood and lymphatic system disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonapegsomatropin/Lonapegsomatropin (N=73) | Placebo/Lonapegsomatropin (N=73) | Somatropin/Lonapegsomatropin (N=74)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 7 (11) | 8 (8)
Nasopharyngitis (Infections and infestations) | 12 (17) | 6 (10) | 2 (2)
Headache (General disorders) | 5 (6) | 5 (5) | 4 (6)
COVID-19 (Infections and infestations) | 4 (4) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 6 (7) | 4 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (11) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 6 (10) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 5 (5) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 4 (8) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 4 (6)
Fatigue (General disorders) | 0 (0) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT05171855/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT05171855/SAP_001.pdf